CLINICAL TRIAL: NCT03772314
Title: Informing Treatment Decisions in the Central Disorders of Hypersomnolence: A Pragmatic Clinical Trial of Modafinil Versus Amphetamines
Brief Title: Modafinil Versus Amphetamines for the Treatment of Narcolepsy Type 2 and Idiopathic Hypersomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Lynn Marie Trotti, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00108167
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Hypersomnia; Narcolepsy Without Cataplexy
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — Modafinil; SLI381; Adderall

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modafinil (Active Comparator): Participants in this study arm will take modafinil.
  Interventions: Drug: Modafinil
- Amphetamine-dextroamphetamine (Experimental): Participants in this study arm will take amphetamine-dextroamphetamine (amphetamine salts).
  Interventions: Drug: Amphetamine-Dextroamphetamine

INTERVENTIONS:
Drug: Modafinil — Participants will received 100-400 milligrams (mg) per day of modafinil for 12 weeks.
  Other Names: Provigil
  Arms: Modafinil
Drug: Amphetamine-Dextroamphetamine — Participants will receive 10-40 mg/day of oral amphetamine salts for 12 weeks.
  Other Names: Adderall
  Arms: Amphetamine-dextroamphetamine

SUMMARY:
For diseases that cause excessive daytime sleepiness (such as narcolepsy and idiopathic hypersomnia), there are several medications that can be used to treat sleepiness. However, it can be difficult to decide which medication to use for a particular individual for several reasons: 1) there are very few studies that directly compare two medications to see which works best; 2) there are very few studies that include people with a disorder of sleepiness called idiopathic hypersomnia.

To address this gap in knowledge, the researchers propose a randomized clinical trial comparing modafinil and amphetamine salts in patients with narcolepsy type 2 or idiopathic hypersomnia. All participants will either receive modafinil or amphetamine salts - no participant will receive placebo.

This study will evaluate which medication works better to improve sleepiness. The researchers will also see which medication is better for other symptoms including difficulty waking up and difficulty thinking, as well as seeing which medication causes fewer side effects. Finally, this study will see if any information about patients (such as age or sleep study features) predicts responding better to one medication or the other.

DETAILED DESCRIPTION:
Currently, there are insufficient data to guide clinical practice regarding the use of amphetamines for the treatment of narcolepsy. This may be particularly important in the case of narcolepsy type 2, for which randomized, controlled trial data show that other treatments are less beneficial than they are for participants with narcolepsy type 1. For the closely related disorder of idiopathic hypersomnia, clinical trial data to guide treatment decision-making are even more limited, with only three published controlled trials ever performed.

To address these evidence gaps, the researchers propose a randomized, active-treatment controlled trial comparing modafinil and amphetamine salts for the treatment of narcolepsy type 2 and idiopathic hypersomnia. The primary outcome will be reduction in excessive daytime sleepiness, as measured by change in Epworth Sleepiness Scale scores from baseline to week 12 on treatment. Other important patient-reported outcomes will be considered as secondary outcomes, including Patient Global Impression of Change for overall severity, sleep inertia, cognitive dysfunction, and sleepiness, as well as other symptom questionnaires.

In addition to directly comparing the efficacy of these two medications for hypersomnolent patients, this study will also evaluate for relatively safety in this population. Further, this study will assess clinical predictors of treatment response. All three of these aims will be complementary in informing shared decision-making about whether to treat with modafinil or amphetamine salts.

Forty-four adult patients seeking evaluation at the Emory Sleep Center for narcolepsy type 2 or idiopathic hypersomnia will be invited to participate and will be randomized to one of the treatment arms upon consent. Participants will receive study treatment for 12 weeks. Participants complete questionnaires at baseline, week 4, week 8, and week 12, with week 12 as the pre-specified primary time point of assessment.

ELIGIBILITY:
Inclusion Criteria:

* narcolepsy type 2 or idiopathic hypersomnia
* ability to give informed consent

Exclusion Criteria:

* contraindication to modafinil or amphetamine salts (history of left ventricular hypertrophy, mitral valve prolapse, other cardiac structural abnormalities, severe cardiovascular disease, unstable angina, myocardial infarction, cardiomyopathy, severe arrhythmias, uncontrolled hypertension, severe hepatic impairment, substance abuse history, psychosis, glaucoma, Tourette's syndrome, and epilepsy)
* obstructive sleep apnea (Apnea-Hypopnea Index (AHI) > 15)
* severe periodic limb movements of sleep with arousals (periodic limb movements (PLM) arousal index > 30)
* allergy to either of the study drugs
* pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Marie Trotti, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Emory Sleep Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trotti LM, Blake T, Hoque R, Rye DB, Sharma S, Bliwise DL. Modafinil Versus Amphetamine-Dextroamphetamine For Idiopathic Hypersomnia and Narcolepsy Type 2: A Randomized, Blinded, Non-inferiority Trial. CNS Drugs. 2024 Nov;38(11):909-920. doi: 10.1007/s40263-024-01122-y. Epub 2024 Sep 21. PMID 39306601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Sleep Center in Atlanta, Georgia, USA. Participant enrollment began April 15, 2019 and all follow-up assessments were completed by April 3, 2023.
Groups:
- Modafinil: Participants with narcolepsy type 2 or idiopathic hypersomnia randomized to take modafinil. Participants received 100-400 milligrams (mg) per day of modafinil for 12 weeks.
- Amphetamine-dextroamphetamine: Participants with narcolepsy type 2 or idiopathic hypersomnia randomized to take amphetamine-dextroamphetamine (amphetamine salts). Participants received 10-40 mg/day of oral amphetamine salts for 12 weeks.
Period: Overall Study
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Started | 22 | 22
Completed | 15 | 20
Not Completed | 7 | 2
Not completed — Adverse Event | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Modafinil: Participants with narcolepsy type 2 or idiopathic hypersomnia randomized to take modafinil. Participants received 100-400 mg/day of modafinil for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Modafinil | Amphetamine-dextroamphetamine | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (8.9) | 35.8 (9.1) | 35.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44
Hypersomnolence diagnosis [Count of Participants; unit: Participants]
  Narcolepsy type 2 (NT2) | 5 | 6 | 11
  Idiopathic hypersomnia (IH), | 17 | 16 | 33
Newly diagnosed at study entry [Count of Participants; unit: Participants] | 17 | 16 | 33
Prior exposure to modafinil [Count of Participants; unit: Participants] | 0 | 1 | 1
Prior exposure to amphetamine-dextroamphetamine [Count of Participants; unit: Participants] | 1 | 2 | 3
Baseline Epworth Sleepiness Scale (ESS) Score [Mean (Standard Deviation); unit: units on a scale] — The ESS asks respondents to indicate how likely they are to doze off or fall asleep during daytime situations such as reading or talking to someone. There are 8 items which are answered on a scale of 0 to 4 where 0 = would never doze and 4 = high chance of dozing. Total score can range from 0 to 24, with higher scores indicating more sleepiness.
  units on a scale | 14.0 (5.3) | 15.2 (3.8) | 14.6 (4.6)
Hypersomnia Severity Index (HSI) Score [Mean (Standard Deviation); unit: score on a scale] — The HSI is a 9-item instrument assessing the severity of excessive sleepiness (hypersomnolence). Items are scored on a Likert scale where 0 = not at all and 4 = very much. Total scores range from 0 to 36 and higher scores indicate greater severity of symptoms of hypersomnia.
  score on a scale | 25.0 (5.9) | 26.5 (6.4) | 25.8 (6.1)
Sleep Inertia Questionnaire (SIQ) Score [Mean (Standard Deviation); unit: score on a scale] — The SIQ is an instrument with 21 items with responses on a 5-point scale where 1 = "not at all" and 5 = "all the time". Two additional questions relate to how much time it takes for the respondent to wake up in the morning. For these analyses, the sum of the 21 items is reported, ranging from 21 to 105, with higher scores indicating increased difficulty with awakening.
  score on a scale | 76.5 (17.5) | 74.0 (13.8) | 75.2 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Epworth Sleepiness Scale (ESS) Score
Description: The Epworth Sleepiness Scale (ESS) asks respondents to indicate how likely they are to doze off or fall asleep during daytime situations such as reading or talking to someone. There are 8 items which are answered on a scale of 0 to 4 where 0 = would never doze and 4 = high chance of dozing. Total score can range from 0 to 24, with higher scores indicating more sleepiness. A score of 0 to 5 can be interpreted as "lower normal daytime sleepiness", a score of 6 to 10 is "higher normal daytime sleepiness", score between 11 to 12 are "mild excessive daytime sleepiness, scores of 13 to 15 are "moderate excessive daytime sleepiness" and scores of 16 to 24 indicate "severe excessive daytime sleepiness". The change in ESS score is obtained by subtracting the total score at week 12 from the baseline score. Scores above 0 mean that the mean score at Week 12 was lower than the mean score at Baseline, indicating less sleepiness.
Time Frame: Baseline, Week 12
Population: This analysis includes the modified intent to treat study population consisting of all participants who were randomized and took at least one dose of study medication. The last observation is used for participants who did not complete the study or had missing responses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 22
score on a scale | 5.0 (2.7) | 4.4 (4.7)

2. Secondary Outcome: Number of Participants Reporting Any Improvement by Patient Global Impression of Change (PGIC) for Overall Disease Severity Score
Description: The PGIC for Overall Severity asks respondents to rate their overall disease compared to baseline. Responses are indicated on a 7-point scale where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". Responses were dichotomized into groups of participants who were treatment responders having any level of improvement (responses of "minimally improved", "much improved", or "very much improved") and treatment non-responders (responses of "no change" to "very much worse"). The number of participants reporting any improvement at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: This analysis includes the modified intent to treat study population consisting of all participants who were randomized and took at least one dose of study medication. The last observation is used for participants who did not complete the study or had missing responses. Two participants in the amphetamine-dextroamphetamine group withdrew prior to completing any PGIC scales and are not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 18 | 16

3. Secondary Outcome: Number of Participants Reporting Much or Very Much Improvement by Patient Global Impression of Change (PGIC) for Overall Disease Severity Score
Description: The PGIC for Overall Severity asks respondents to rate their overall disease compared to baseline. Responses are indicated on a scale of 1 to 7 where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". The number of participants reporting "much improved" or "very much improved" at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 13 | 10

4. Secondary Outcome: Number of Participants Reporting Any Improvement From Baseline on Patient Global Impression of Change (PGIC) for Sleepiness Score
Description: The PGIC for Sleepiness asks respondents to rate their sleepiness compared to baseline. Responses are indicated on a 7-point scale where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". Responses were dichotomized into groups of participants who were treatment responders having any level of improvement (responses of "minimally improved", "much improved", or "very much improved") and treatment non-responders (responses of "no change" to "very much worse"). The number of participants reporting any improvement at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 19 | 16

5. Secondary Outcome: Number of Participants Reporting Much or Very Much Improvement From Baseline on Patient Global Impression of Change (PGIC) for Sleepiness Score
Description: The PGIC for Sleepiness asks respondents to rate their sleepiness compared to baseline. Responses are indicated on a 7-point scale where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". The number of participants reporting "much improved" or "very much improved" at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 14 | 10

6. Secondary Outcome: Number of Participants Reporting Any Improvement With Patient Global Impression of Change (PGIC) for Cognitive Dysfunction Score
Description: The PGIC for Cognitive Dysfunction asks respondents to rate their cognitive dysfunction compared to baseline. Cognitive dysfunction is defined for participants as "difficulty with thinking, problems with attention or concentration, and/or brain fog". Responses are indicated on a scale of 1 to 7 where where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". Responses were dichotomized into groups of participants who were treatment responders having any level of improvement (responses of "minimally improved", "much improved", or "very much improved") and treatment non-responders (responses of "no change" to "very much worse"). The number of participants reporting any improvement at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 16 | 13

7. Secondary Outcome: Number of Participants Reporting Much or Very Much Improvement With Patient Global Impression of Change (PGIC) for Cognitive Dysfunction Score
Description: The PGIC for Cognitive Dysfunction asks respondents to rate their cognitive dysfunction compared to baseline. Cognitive dysfunction is defined for participants as "difficulty with thinking, problems with attention or concentration, and/or brain fog". Responses are indicated on a scale of 1 to 7 where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". The number of participants reporting "much improved" or "very much improved" at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 5 | 10

8. Secondary Outcome: Number of Participants Reporting Any Improvement by Patient Global Impression of Change (PGIC) for Sleep Inertia Score
Description: The PGIC for Sleep Inertia asks respondents to rate their sleep inertia compared to baseline. Sleep inertia is defined for participants as "difficulty waking up and getting out of bed in the morning because of sleepiness". Responses are indicated on a scale of 1 to 7 where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". Responses were dichotomized into groups of participants who were treatment responders having any level of improvement (responses of "minimally improved", "much improved", or "very much improved") and treatment non-responders (responses of "no change" to "very much worse"). The number of participants reporting any improvement at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 11 | 11

9. Secondary Outcome: Number of Participants Reporting Much or Very Much Improvement by Patient Global Impression of Change (PGIC) for Sleep Inertia Score
Description: The PGIC for Sleep Inertia asks respondents to rate their sleep inertia compared to baseline. Sleep inertia is defined for participants as "difficulty waking up and getting out of bed in the morning because of sleepiness". Responses are indicated on a scale of 1 to 7 where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved" 4 = "no change", 5 = "minimally worse", 6 = "much worse" and 7 = "very much worse". The number of participants reporting "much improved" or "very much improved" at the Week 12 assessment compared to how they felt right before starting the study medication was examined.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 20
Participants | 4 | 4

10. Secondary Outcome: Change in Hypersomnia Severity Index (HSI) From Baseline
Description: The HSI is a 9-item instrument assessing the severity of excessive sleepiness (hypersomnolence). Items are scored on a Likert scale where 0 = not at all and 4 = very much. Total scores range from 0 to 36 and higher scores indicate greater severity of symptoms of hypersomnia. The change in HSI score is obtained by subtracting the total score at week 12 from the baseline score. Scores above 0 signify that the mean score at Week 12 was lower than the mean score at Baseline, indicating reduced severity of hypersomnia symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 22
score on a scale | 8.0 (5.6) | 10.4 (6.8)

11. Secondary Outcome: Change in Sleep Inertia Questionnaire (SIQ) Score From Baseline
Description: The SIQ is an instrument with 21 items with responses on a 5-point scale where 1 = "not at all" and 5 = "all the time". Two additional questions relate to how much time it takes for the respondent to wake up in the morning. For these analyses, a total score for the 21 items was generated. The change in SIQ score is obtained by subtracting the total score at week 12 from the baseline score. Scores above 0 signify that the mean score at Week 12 was lower than the mean score at Baseline, indicating reduced difficulty awakening.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
Number analyzed (Participants) | 22 | 22
score on a scale | 19.0 (15.9) | 18.2 (18.4)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected once participants began taking the study medication and continued through the final assessment at Week 12.
Description: Only treatment-emergent adverse events were collected for this study.
Arm/Group | Modafinil | Amphetamine-dextroamphetamine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 17/22 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil (N=22) | Amphetamine-dextroamphetamine (N=22)
Hospitalization due to suicidal ideation (Psychiatric disorders) | 1 | 0 — The participant's psychiatric team continued the study medication and symptoms were successfully managed.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil (N=22) | Amphetamine-dextroamphetamine (N=22)
Reduced appetite (General disorders) | 2 | 8
Headache (General disorders) | 4 | 6
Insomnia (General disorders) | 5 | 3
Anxiety symptoms (Psychiatric disorders) | 5 | 0
Dizziness (General disorders) | 1 | 4
Elevated heart rate/palpitations (Cardiac disorders) | 2 | 2
Jitteriness (General disorders) | 2 | 2
Depressive symptoms (Psychiatric disorders) | 3 | 1
Nausea (General disorders) | 3 | 1
Dry mouth (General disorders) | 1 | 3
Elevated blood pressure (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT03772314/Prot_SAP_000.pdf